CLINICAL TRIAL: NCT02012790
Title: Clinical & Metabolic Effects of Altering n-3 & n-6 Fatty Acids in Migraine (RCT)
Brief Title: Nutrition for Migraine Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-3284; UL1TR000083 (NIH); 1R01AT007813-01A1 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-12-16 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Migraine Disorders
Keywords: Migraine disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet A (Experimental): Whole food diet modifies dietary fatty acids. Foods provided for 16 weeks; study oils provided for 22 weeks.
  Interventions: Other: Diet
- Diet B (Experimental): Whole food diet modifies dietary fatty acids. Foods provided for 16 weeks; study oils provided for 22 weeks.
  Interventions: Other: Diet
- Diet C (Active Comparator): Whole food diet modifies dietary fatty acids. Foods provided for 16 weeks; study oils provided for 22 weeks.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — The dietary intervention provides dietary counseling, whole foods (enough for 2 meals and 2 snacks per day) including study oils

SUMMARY:
Migraine is a widespread, debilitating, chronic pain disorder and a major public health challenge. Most conventional, pharmaceutical treatments fail to give satisfactory long-term relief and their repeated use can have important side effects. This project involves implementation of substantial dietary changes in adults with migraine. Our goal is to test the hypothesis that a causal relationship exists between migraine symptoms and the amount and proportions of foods consumed containing defined amounts of polyunsaturated fatty acids.

Significant findings supporting the hypothesis will lead to a major shift in both prevention and management of migraine and other chronic pain disorders. Emphasis is on low-cost, health improvement strategies utilizing specific dietary modifications for pain management, based on solid clinical research evidence.

DETAILED DESCRIPTION:
Episodic migraine is a debilitating chronic pain condition afflicting 12% of American adults. Current conventional treatments rely on medications that provide limited or transient relief, target symptoms rather than the underlying causes of pain, and are associated with significant side effects and costs. It is therefore essential to investigate non-pharmacologic approaches to conventional headache treatments. Certain fatty acids and their bioactive metabolites regulate multiple pain-related biochemical pathways. Controlled clinical trials investigating pain modulation in response to dietary changes while exploring relevant mechanisms of action in humans are lacking.

In a recent feasibility study in patients with chronic daily headache (CDH), we found that targeted fatty acid modifications altered circulating endovanilloids, while reducing headache frequency and improving quality of life. These findings support our proposed model in which diet-induced alterations in endovanilloids modulate transient receptor potential cation channel subfamily V member 1 (TRPV1) activity in vivo, leading to important implications for migraine and chronic pain in general.

The goal of this research is to assess whether dietary PUFA modifications can result in predicted changes in circulating endovanilloids and improvement in headache-related clinical outcomes. The proposed 3-arm, 26-week,randomized, controlled, single-blind trial, with 51 subjects in each group, includes a 4-week baseline of usual care, followed by randomization to one of three 22-week dietary interventions plus usual care. Each of the three arms involves specific modifications of dietary fatty acid intakes through a whole foods diet. Participants in the dietary interventions receive food sufficient for 2 meals and 2 snacks daily along with extensive dietary counseling.

Specific aims are:

1. To assess the efficacy of the dietary interventions in inducing the predicted changes in circulating fatty acid endovanilloid derivatives;
2. To compare the clinical effects in migraine specific outcomes of two 16-week analgesic dietary interventions with each other and a control diet;
3. To test, in an exploratory manner, our model of the proposed causal chain linking changes in fatty acids, their endovanilloid derivatives, and headache clinical endpoints.

This proposal utilizes an innovative design and hypotheses to address current research funding priorities, by examining clinical efficacy and underlying mechanisms of a promising dietary manipulation with the distinct potential for high impact in terms of ameliorating a chronic, disabling pain disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Either gender
* Meets 2004 International Classification of Headache Disorders-II* criteria for Episodic Migraine
* Frequent migraine headaches
* Headache history: > 2 years leading up to study meeting migraine criteria
* Willing to complete daily diary for 26 weeks
* Able to attend 8 dietitian counseling sessions
* Under care of a physician for headaches
* Able to read and communicate in English

Exclusion Criteria:

* Marked depression, anxiety or psychosis.
* History of specific food allergies, such as, but not limited to, dairy or gluten products
* Pregnancy or anticipated pregnancy
* Active treatment for a major medical illness, such as malignancy, autoimmune, immune deficiency disorder, etc.
* History of significant head trauma or head/neck surgery within the past 3 years
* History of subarachnoid or intra-cerebral hemorrhage or subdural hematoma
* Allergy to fish or strong aversion to fish consumption.
* History of nervous system infection such as meningitis or encephalitis within the preceding 5 years
* History of vasculitis, intracranial mass, clotting disorder
* Cognitive dysfunction that would prevent informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-07; Primary Completion 2018-03-29 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Primary metabolic outcome: 17-hydroxy docosahexaenoic acid (DHA) | Change in 17-hydroxy DHA at 16 weeks
  17-hydroxy DHA is the pathway marker and precursor to two families of potent bioactive mediators with analgesic properties (D series resolvins and protectins), which will be measured at baseline and after 16 weeks of diet exposure.
Primary clinical outcome: Headache-specific Quality of Life (HIT-6) | Change in HIT-6 at 16 weeks
  The HIT-6 is a validated questionnaire designed "to measure the impact that headaches have on the ability to function on the job, at school, at home, and in social situations"

SECONDARY OUTCOMES:
Headache hours per day (headache frequency) are measured by a daily Headache Diary | Trajectory of change: -4 to 0 weeks (pre-intervention), 0-16 weeks (intervention), and 16-22 weeks (post-intervention)
  Subjects will be instructed to maintain a daily record of their headaches using a headache diary. Subjects will be asked to record the frequency, intensity, and duration of their headaches by rating their headaches hourly as "none", "mild", "moderate" and "severe". Hours of sleep will also be indicated. In our clinical trial of a migraine headache treatment, subjects were willing and able to complete daily diaries with minimal loss of data. Diaries will be completed on a secure website via a computer or smart-phone interface. Numbers of hours of any headache will be calculated along with numbers of hours of moderate to severe headache for use in longitudinal models.
Patient-Reported Outcomes Measurement Information System-29 Profile | Pre-post and trajectory of change measured at randomization and at 4,10, and 16 weeks after randomization
  This battery of short instruments covers the following domains associated with chronic pain: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with social role, pain interference, and pain intensity
17-hydroxy DHA trajectory | Trajectory of change in 17-hydroxy DHA 0-16 weeks and 16-22 weeks
  17-hydroxy DHA is the pathway marker and precursor to two families of potent bioactive mediators with analgesic properties (D series resolvins and protectins), which will be measured at baseline, after 4, 10, and 16 weeks of diet exposure, and at the end of the observation period (22 weeks).
HIT-6 | Trajectory of change pre-intervention, 0-16 weeks, and 16-22 weeks
  The HIT-6 is a validated questionnaire designed "to measure the impact that headaches have on the ability to function on the job, at school, at home, and in social situations" measured at baseline, randomization, and after 4,10, and 16 weeks on the diet and at the end of the observation period (22 weeks)

OTHER OUTCOMES:
Migraine Disability Assessment Score (MIDAS) | Change in MIDAS from randomization to 16 weeks after randomization
  Disability, defined as the consequences of illness on ability to work and function, will be measured using the headache disability assessment score (MIDAS). Derived from the Headache Impact Test, MIDAS is a 7-item questionnaire that assesses the number of days during the previous three months that respondents missed work or school, experienced decreased productivity at work or home, or missed social engagements because of headaches. Test-retest reliability is acceptable, with Spearman's correlation coefficient ranging from 0.67 to 0.73. Cronbach's alpha is 0.83
Medication use for treatment of headache. | trajectory of change over 16 weeks
  Subjects enter number of doses of medications used for treatment of headaches into their daily diaries.
Unusual symptoms | Daily for 4 weeks before randomization, and 22 weeks after randomization
  Subjects will record unusual symptoms in a comment field in their daily diaries.

CONTACTS AND LOCATIONS:
Overall Officials: John D Mann, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Program on Integrative Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Faurot KR, Park J, Miller V, Honvoh G, Domeniciello A, Mann JD, Gaylord SA, Lynch CE, Palsson O, Ramsden CE, MacIntosh BA, Horowitz M, Zamora D. Dietary fatty acids improve perceived sleep quality, stress, and health in migraine: a secondary analysis of a randomized controlled trial. Front Pain Res (Lausanne). 2023 Oct 25;4:1231054. doi: 10.3389/fpain.2023.1231054. eCollection 2023. PMID 37954068
- [Derived] Ramsden CE, Zamora D, Faurot KR, MacIntosh B, Horowitz M, Keyes GS, Yuan ZX, Miller V, Lynch C, Honvoh G, Park J, Levy R, Domenichiello AF, Johnston A, Majchrzak-Hong S, Hibbeln JR, Barrow DA, Loewke J, Davis JM, Mannes A, Palsson OS, Suchindran CM, Gaylord SA, Mann JD. Dietary alteration of n-3 and n-6 fatty acids for headache reduction in adults with migraine: randomized controlled trial. BMJ. 2021 Jun 30;374:n1448. doi: 10.1136/bmj.n1448. PMID 34526307
- [Derived] Miller VE, Faurot KR, Palssson OS, MacIntosh BA, Suchindran C, Honvoh G, Gaylord S, Ramsden CE, Mann JD. Comparing prospective headache diary and retrospective four-week headache questionnaire over 20 weeks: Secondary data analysis from a randomized controlled trial. Cephalalgia. 2020 Nov;40(13):1523-1531. doi: 10.1177/0333102420949180. Epub 2020 Aug 16. PMID 32799667
- [Derived] Mann JD, Faurot KR, MacIntosh B, Palsson OS, Suchindran CM, Gaylord SA, Lynch C, Johnston A, Maiden K, Barrow DA, Hibbeln JR, Ramsden CE. A sixteen-week three-armed, randomized, controlled trial investigating clinical and biochemical effects of targeted alterations in dietary linoleic acid and n-3 EPA+DHA in adults with episodic migraine: Study protocol. Prostaglandins Leukot Essent Fatty Acids. 2018 Jan;128:41-52. doi: 10.1016/j.plefa.2017.11.002. Epub 2017 Nov 16. PMID 29413360